CLINICAL TRIAL: NCT03094156
Title: A Double-blind, Randomised, Placebo-controlled, Rising Multiple Dose Study in Healthy Volunteers to Investigate the Effect of BIA 6-512 at Steady-state on the Levodopa Pharmacokinetics When Administered in Combination With a Single-dose of Levodopa/Benserazide 200/50 mg or With a Single-dose of Levodopa/Benserazide 200/50 mg Plus a Single-dose of Entacapone 200 mg
Brief Title: Effect of BIA 6-512 at Steady-state on the Levodopa Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: BIA-6512-106
Record Dates: First submitted 2017-03-23; First posted 2017-03-29 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Resveratrol; entacapone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo (Experimental): Subjects were administered with those investigational products at approximately 8-h intervals, starting in the morning (approximately at 8h00) of Day 1 and finishing in the morning of Day 5 (last dose). On Day 4, concomitantly with the Placebo morning dose, one tablet of Madopar® 250 was administered. On Day 5, concomitantly with the Placebo morning dose, one tablet of Madopar® 250 and one tablet of Comtan® were administered.
  Interventions: Drug: Placebo; Drug: Madopar® 250; Drug: Comtan®
- BIA 6-512 25 mg (Experimental): Subjects were administered with those investigational products at approximately 8-h intervals, starting in the morning (approximately at 8h00) of Day 1 and finishing in the morning of Day 5 (last dose). On Day 4, concomitantly with the BIA 6-512 25 mg morning dose, one tablet of Madopar® 250 was administered. On Day 5, concomitantly with the BIA 6-512 25 mg morning dose, one tablet of Madopar® 250 and one tablet of Comtan® were administered.
  Interventions: Drug: BIA 6-512; Drug: Madopar® 250; Drug: Comtan®
- BIA 6-512 50 mg (Experimental): Subjects were administered with those investigational products at approximately 8-h intervals, starting in the morning (approximately at 8h00) of Day 1 and finishing in the morning of Day 5 (last dose). On Day 4, concomitantly with the BIA 6-512 50 mg morning dose, one tablet of Madopar® 250 was administered. On Day 5, concomitantly with the BIA 6-512 50 mg morning dose, one tablet of Madopar® 250 and one tablet of Comtan® were administered.
  Interventions: Drug: BIA 6-512; Drug: Madopar® 250; Drug: Comtan®
- BIA 6-512 75 mg (Experimental): Subjects were administered with those investigational products at approximately 8-h intervals, starting in the morning (approximately at 8h00) of Day 1 and finishing in the morning of Day 5 (last dose). On Day 4, concomitantly with the BIA 6-512 75 mg morning dose, one tablet of Madopar® 250 was administered. On Day 5, concomitantly with the BIA 6-512 75 mg morning dose, one tablet of Madopar® 250 and one tablet of Comtan® were administered.
  Interventions: Drug: BIA 6-512; Drug: Madopar® 250; Drug: Comtan®
- BIA 6-512 100 mg (Experimental): Subjects were administered with those investigational products at approximately 8-h intervals, starting in the morning (approximately at 8h00) of Day 1 and finishing in the morning of Day 5 (last dose). On Day 4, concomitantly with the BIA 6-512 100 mg morning dose, one tablet of Madopar® 250 was administered. On Day 5, concomitantly with the BIA 6-512 100 mg morning dose, one tablet of Madopar® 250 and one tablet of Comtan® were administered.
  Interventions: Drug: BIA 6-512; Drug: Madopar® 250; Drug: Comtan®

INTERVENTIONS:
Drug: Placebo — 1 capsule of placebo [to be taken orally, with 240 mL of potable water]
  Arms: Placebo
Drug: BIA 6-512 — 1 capsule of BIA 6-512 25mg or 1 capsule of BIA 6-512 50 mg or 1 capsule of BIA 6-512 75 mg or 1 capsule of BIA 6-512 100 mg [to be taken orally, with 240 mL of potable water]
  Other Names: Trans-resveratrol
  Arms: BIA 6-512 100 mg; BIA 6-512 25 mg; BIA 6-512 50 mg; BIA 6-512 75 mg
Drug: Madopar® 250 — Levodopa/benserazide immediate release tablets 200mg/50mg [to be taken orally, with 240 mL of potable water]
Drug: Comtan® — Entacapone 200 mg tablets [to be taken orally, with 240 mL of potable water]

SUMMARY:
The purpose of the study was to To investigate whether the administration of BIA 6-512 (25 mg, 50 mg, 75 mg and 100 mg) at steady-state affects the pharmacokinetics of levodopa when administered in combination with a single-dose of immediate release levodopa/benserazide 200/50 mg or with a single-dose of immediate release levodopa/benserazide 200/50 mg plus a single-dose of entacapone 200 mg.

DETAILED DESCRIPTION:
Single centre, double-blind, randomised, placebo-controlled, rising multiple-dose study in four sequential groups of healthy male and female subjects. Eligible subjects were admitted to the Human Pharmacology Unit (UFHBIAL - Portela & Cª, SA) on the day prior to receiving the first study medication. Starting in the morning of Day 1 (first dose), subjects received BIA 6-512/Placebo thrice-daily until the morning of Day 5 (last dose). Concomitantly with the morning dose of BIA 6-512/Placebo, on Day 4 a levodopa/benserazide 200/50 mg (Madopar® 250) single-dose was administered. On Day 5, a Madopar® 250 single-dose and a entacapone 200 mg (Comtan®) single-dose were administered concomitantly with the morning dose of BIA 6-512/Placebo. In the morning of Day 4 and Day 5, products were administered in fasting of at least 8 hours and subjects remained fasted until 2 h post-dose. Subjects were resident in the UFH from admission (Day 0) until at least 24 h post last dose (Day 6); then, they were discharged and returned for the follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged between 18 and 45 years, inclusive.
* Subjects of body mass index (BMI) between 19 and 30 kg/m2, inclusive.
* Subjects who were healthy as determined by pre-study medical history, physical examination, vital signs, complete neurological examination and 12-lead ECG.
* Subjects who had negative tests for HBsAg, anti-HCVAb and HIV-1 and HIV-2 Ab at screening
* Subjects who had clinical laboratory test results clinically acceptable at screening and admission.
* Subjects who had a negative screen for alcohol and drugs of abuse at screening and admission.
* Subjects who were non-smokers or who smoked ≤ 10 cigarettes or equivalent per day.
* Subjects who were able and willing to gave written informed consent.
* (If female) She was not of childbearing potential by reason of surgery or, if of childbearing potential, she used one of the following methods of contraception: double barrier, intrauterine device or abstinence.
* (If female) She had a negative urine pregnancy test at screening and admission.

Exclusion Criteria:

* Subjects who had a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders.
* Subjects who had a clinically relevant surgical history.
* Subjects who had a clinically relevant family history.
* Subjects who had a history of relevant atopy.
* Subjects who had a history of relevant drug hypersensitivity.
* Subjects who had a history of alcoholism or drug abuse.
* Subjects who consumed more than 14 units of alcohol a week.
* Subjects who had a significant infection or known inflammatory process on screening or admission.
* Subjects who had acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhoea, heartburn) at the time of screening or admission.
* Subjects who had used medicines within 2 weeks of admission that may affect the safety or other study assessments, in the investigator's opinion.
* Subjects who had previously participated in a clinical trial with BIA 6-512.
* Subjects who had used any investigational drug or participated in any clinical trial within 6 months prior to screening.
* Subjects who had participated in more than 2 clinical trials within the 12 months prior to screening.
* Subjects who had donated or received any blood or blood products within the 3 months prior to screening.
* Subjects who were vegetarians, vegans or have medical dietary restrictions.
* Subjects who cannot communicate reliably with the investigator.
* Subjects who were unlikely to co-operate with the requirements of the study.
* Subjects who were unwilling or unable to give written informed consent.
* (If female) She was pregnant or breast-feeding.
* (If female) She was of childbearing potential and she did not use an effective contraceptive method (double-barrier, intra-uterine device or abstinence) or she used oral contraceptives.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2006-04-26 (Actual); Primary Completion 2006-07-11 (Actual); Study Completion 2006-07-11 (Actual)

PRIMARY OUTCOMES:
Day 4 - Maximum observed plasma drug concentration (Cmax) | pre-dose, ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8 and 16 hours post-dose
  BIA 6-512, levodopa, 3-OMD and entacapone pharmacokinetic parameters on day 4
Day 4 - Time of occurrence of Cmax (tmax) | pre-dose, ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8 and 16 hours post-dose
  BIA 6-512, levodopa, 3-OMD and entacapone pharmacokinetic parameters on day 4
Day 4 - Area under the plasma concentration-time curve (AUC) from time zero to the last sampling time at which concentrations were at or above the limit of quantification (AUC0-t) | pre-dose, ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8 and 16 hours post-dose
  BIA 6-512, levodopa, 3-OMD and entacapone pharmacokinetic parameters on day 4
Day 4 - AUC from time zero to 8 h post-dose (AUC0-τ) | pre-dose, ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8 and 16 hours post-dose
  BIA 6-512, levodopa, 3-OMD and entacapone pharmacokinetic parameters on day 4
Day 4 - Apparent terminal elimination half-life, calculated from ln 2/λz (t1/2) | pre-dose, ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8 and 16 hours post-dose
  BIA 6-512, levodopa, 3-OMD and entacapone pharmacokinetic parameters on day 4
Day 4 - Area under the plasma concentration versus time curve from time zero to infinity (AUC0-∞) | pre-dose, ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8 and 16 hours post-dose
  BIA 6-512, levodopa, 3-OMD and entacapone pharmacokinetic parameters on day 4
Day 5 - Maximum observed plasma drug concentration (Cmax) | pre-dose, ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 16 and 24 hours post-dose
Day 5 - Time of occurrence of Cmax (tmax) | pre-dose, ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 16 and 24 hours post-dose
  BIA 6-512, levodopa, 3-OMD and entacapone pharmacokinetic parameters on day 5
Day 5 - Area under the plasma concentration-time curve (AUC) from time zero to the last sampling time at which concentrations were at or above the limit of quantification (AUC0-t) | pre-dose, ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 16 and 24 hours post-dose
  BIA 6-512, levodopa, 3-OMD and entacapone pharmacokinetic parameters on day 5
Day 5 - AUC from time zero to 8 h post-dose (AUC0-τ) | pre-dose, ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 16 and 24 hours post-dose
  BIA 6-512, levodopa, 3-OMD and entacapone pharmacokinetic parameters on day 5
Day 5 - Apparent terminal elimination half-life, calculated from ln 2/λz (t1/2) | pre-dose, ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 16 and 24 hours post-dose
  BIA 6-512, levodopa, 3-OMD and entacapone pharmacokinetic parameters on day 5
Day 5 - Area under the plasma concentration versus time curve from time zero to infinity (AUC0-∞) | pre-dose, ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 16 and 24 hours post-dose
  BIA 6-512, levodopa, 3-OMD and entacapone pharmacokinetic parameters on day 5

CONTACTS AND LOCATIONS:
Locations (1):
- Human Pharmacology Unit (UFH) - BIAL - Portela & Cª, SA, S. Mamede Do Coronado, Portugal

IPD SHARING:
Plan to Share IPD: Undecided